CLINICAL TRIAL: NCT02341079
Title: Prospective Randomized Trial Comparing Intraoperative Liposomal Bupivacaine Injection With Indwelling Femoral Nerve Blockade in Early Postoperative Pain Control for Primary Total Knee Arthroplasty
Brief Title: Intraoperative Liposomal Bupivacaine Injection in Primary Total Knee Arthroplasty
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Principal no longer interested in conducting study
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD.2014.0101
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee; Arthritis, Degenerative; Osteoarthrosis; Osteoarthrosis Deformans
Keywords: Total Knee Arthroplasty; Osteoarthritis; Femoral Nerve Blockade; Liposomal Bupivacaine
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femoral Nerve Blockade (Active Comparator): Femoral nerve block delivered via indwelling femoral nerve catheter
  Interventions: Drug: Indwelling femoral nerve block
- Bupivacaine Liposome Injection (Experimental): Intraoperative intracapsular injection of bupivacaine liposome
  Interventions: Drug: Bupivacaine Liposome Injection

INTERVENTIONS:
Drug: Bupivacaine Liposome Injection — Intraoperative intracapsular injection of 266mg of bupivacaine liposome injection diluted to 60mL with 0.9% normal saline.
  Other Names: EXPAREL
  Arms: Bupivacaine Liposome Injection
Drug: Indwelling femoral nerve block — Femoral nerve block delivered via indwelling femoral nerve catheter with 0.125% bupivacaine.
  Arms: Femoral Nerve Blockade

SUMMARY:
The purpose of the study is to evaluate the efficacy of local infiltration of liposomal bupivacaine versus use of an indwelling femoral peripheral nerve block in controlling early postoperative pain in primary total knee arthroplasty. The investigators hope to demonstrate equivalency of treatment modalities to provide an alternative to the commonly used treatment of femoral nerve blockade.

DETAILED DESCRIPTION:
Postoperative pain control in total knee arthroplasty is generally managed by a multimodal approach of premedication, epidural and/or peripheral nerve blocks, narcotic medications, and anti-inflammatories. Multiple studies have evaluated the efficacy of anesthetic "cocktails" of various medications for local tissue infiltration to aide in controlling postoperative pain. A recent systematic review supported the use of local anesthetic infiltration in a single intraoperative dose as an adjunct to femoral nerve block in the relief of pain; with combinations of ropivacaine, ketorolac, and adrenaline providing the best results. Several studies noted decreases in opioid consumption and overall pain scores in the perioperative period.

A novel compound, liposomal bupivacaine (EXPAREL®, Pacira Pharmaceuticals, Inc., Parsippany, NJ, USA), has been proposed for use in total knee arthroplasty. To our knowledge, only one randomized controlled trial involving use of this compound in total knee arthroplasty has been published and was performed as a phase two dose ranging trial comparing liposomal bupivacaine to bupivacaine HCl. No statistically significant difference between the two compounds was shown, but a trend towards benefit in short term pain control was shown with EXPAREL 532mg.

Our current pain management regimen utilizes the multimodal approach of neuraxial anesthesia, indwelling femoral nerve catheter, opioids, and anti-inflammatory medications. The regional anesthesia service manages postoperative pain while the indwelling femoral nerve catheter is in place. The epidural is utilized for early postoperative analgesia and thromboprophylaxis. The epidural is discontinued on post-operative day 1 and the femoral nerve catheter is removed by the morning of postoperative day 3. Although femoral nerve catheters provide excellent pain control following TKA, there are associated disadvantages. Most notably there is inherent quadriceps weakness which places the patient at increased fall risk. To reduce the risk of falling, patients must wear a knee immobilizer with ambulation until the catheter is removed and quadriceps function has returned. This may delay the ability to actively participate in physical therapy.

The purpose of our present study is to evaluate the efficacy of local infiltration of liposomal bupivacaine versus use of an indwelling femoral peripheral nerve block in controlling early postoperative pain. The investigators aim to show equivalency between the two treatment modalities. Our hypothesis is that a systematic local infiltration of liposomal bupivacaine provided intraoperatively is equally efficacious as femoral indwelling peripheral nerve blockade in immediate postoperative pain control with more rapid progression with physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Undergoing unilateral primary total knee arthroplasty

Exclusion Criteria:

* Revision total knee arthroplasty
* Bilateral total knee arthroplasty
* Prior allergy or adverse reaction to local anesthetic
* Hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Pain Scale | 0-3 months
  10cm VAS scale completed by the patient at set intervals postoperatively
Oral and Intravenous Opioid Consumption | 0-5 days (during hospitalization)
  Oral and intravenous opioid use calculated in terms of morphine equivalents
Hospital for Special Surgery (HSS) Knee Scores | 0-3 months
  Standardized functional clinical score for knee symptoms

SECONDARY OUTCOMES:
Length of Hospital Stay | 0-5 days
Distance ambulated with physical therapy | 0-5 days (during hospitalization)
Time to straight leg raise with physical therapy | 0-5 days (during hospitalization)
  Time to return of quadriceps function
Postoperative range of motion | 0-3 months
  Knee range of motion measure by physical therapy and in clinic
Postoperative complication rate | 0-3 months
  All intervention related complications for each arm of the study
Plasma bupivacaine concentrations | 0-5 days (during hospitalization)
  Plasma levels of bupivacaine monitored throughout hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Patrick B Morrissey, M.D., Principal Investigator — Naval Medical Center San Diego Department of Orthopadic Surgery
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States